CLINICAL TRIAL: NCT07281313
Title: High-intensity Exercise in Stroke Recovery: Randomized Trial
Brief Title: Aphasia Physical EXercise Study: Randomized Trial
Acronym: APEX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Collaborators: University of California, San Francisco (Other); California State University, East Bay (Other); University of San Francisco (Other); National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Maria Ivanova, Associate Professional Researcher, University of California, Berkeley
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20243771; R01DC022663 (NIH)
Record Dates: First submitted 2025-11-25; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Aphasia, Acquired; Aphasia; Aphasia, Fluent; Aphasia, Non-fluent; Aphasia Following Cerebral Infarction; Aphasia Following Nontraumatic Intracerebral Hemorrhage
Keywords: aphasia; physical exercise; high intensity interval training; cognition; physical fitness; balance; stroke; language
MeSH Terms: conditions — Aphasia; Aphasia, Wernicke; Aphasia, Broca; Motor Activity; Stroke; Language

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to the low intensity intervention (control intervention) or the high-intensity physical exercise intervention (target intervention).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-intensity physical exercise (Experimental): The participants will take part in a high-intensity Aphasia Physical EXercise (APEX) intervention designed specifically for individuals with chronic post-stroke aphasia for 12 weeks.
  Interventions: Behavioral: High-intensity physical exercise
- Low-intensity physical exercise (Active Comparator): The participants will participate in a low-intensity non-aerobic exercise program for 12 weeks.
  Interventions: Behavioral: Low-intensity physical exercise

INTERVENTIONS:
Behavioral: High-intensity physical exercise — We have developed a new exercise program specifically designed for individuals with post-stroke aphasia, Aphasia Physical EXercise (APEX), to provide a safe, stroke- and aphasia-friendly physical exercise intervention to achieve optimal physical fitness and cognitive/language gains. This intervention, based on published research and clinical practice recommendations, is a high-intensity interval training full-body workout optimized to accommodate the range of motor abilities and general deconditioning observed in stroke survivors.
  Arms: High-intensity physical exercise
Behavioral: Low-intensity physical exercise — As an active control intervention, a low-intensity non-aerobic exercise program was selected that mirrors more closely the standard-of-care physical therapy currently provided to stroke patients. This control intervention will offer the same level of participant involvement and type of interaction, but without the intensity element, i.e., it will not incorporate the cardiovascular and the strengthening components.
  Arms: Low-intensity physical exercise

SUMMARY:
The goal of this clinical trial is to evaluate the effects of a high-intensity exercise program on recovery in individuals with post-stroke aphasia. The high-intensity exercise program has been specifically designed for individuals with post-stroke aphasia and includes an interval training full-body workout, which can increase cardiovascular fitness, improve muscle strength and motor performance, and maximize cognitive and language gains. The main question this study aims to answer is:

• Does participation in a high-intensity exercise program lead to changes in physical health, language, cognitive, motor recovery, psychological and/or psychosocial domains?

Participants will be randomly assigned to either a high-intensity exercise program (target intervention) or a low-intensity exercise program (control intervention) delivered over 12-weeks in a group setting.

Outcome measures will be collected once immediately after the intervention period and once during the following 12-week maintenance period to capture short- and long-term effects of the exercise program.

ELIGIBILITY:
Inclusion Criteria:

* Aphasia following ischemic or hemorrhagic stroke
* Aphasia as determined by a standardized language test (Western Aphasia Battery Aphasia Quotient < 93.8 at study intake)
* At least 6 months from the last stroke
* Proficient in English before the stroke
* At least 8 years of education
* Between the ages of 18 and 80
* Independent with ambulation without a device (single-point cane accepted)
* Medically stable with no contraindications to participate in regular physical exercise as determined by the patients' own primary care provider or other treating provider.

Exclusion Criteria:

* Prior history of dementia, neurologic illness (other than stroke), or recent (last 3 years) substance abuse
* Significant visual or hearing disabilities (e.g., neglect, uncorrected visual or hearing loss) that interfere with testing
* Self-report uncontrolled cardiorespiratory and/or metabolic disorders incompatible with exercise

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2030-10-31 (Estimated); Study Completion 2030-10-31 (Estimated)

PRIMARY OUTCOMES:
Change on the Western Aphasia Battery (WAB) - Aphasia Quotient | (T1) Baseline: at the start of the study; (T2) Pre-treatment: 1 week prior to the start of the intervention; (T3) Post-treatment: the week immediately following the intervention; (T4) Follow-up: 3 months after the conclusion of the intervention.
  The Aphasia Quotient from the Western Aphasia Battery (a standardized language test) measures overall severity of language impairment in aphasia and ranges from 0 to 100, with lower scores indicative of more severe aphasia.

SECONDARY OUTCOMES:
Change on the WAB subtest scores | (T1) Baseline: at the start of the study; (T2) Pre-treatment: 1 week prior to the start of the intervention; (T3) Post-treatment: the week immediately following the intervention; (T4) Follow-up: 3 months after the conclusion of the intervention.
  The subtests from the Western Aphasia Battery (a standardized language test) measure different language capacities. Specifically, we will look at Spontaneous Speech, Fluency, Auditory Verbal Comprehension, Repetition, Naming and Word Finding subtest scores.
Change on the Curtiss-Yamada Comprehensive Language Evaluation - Revised (CYCLE-R) | (T1) Baseline: at the start of the study; (T2) Pre-treatment: 1 week prior to the start of the intervention; (T3) Post-treatment: the week immediately following the intervention; (T4) Follow-up: 3 months after the conclusion of the intervention.
  A sentence-to-picture matching tasks that evaluates comprehension of sentences of varying complexity. The scores range from 0 to 100%, with higher scores indicative of better comprehension abilities.
Changes on Category and Letter Verbal Fluency tasks | (T1) Baseline: at the start of the study; (T2) Pre-treatment: 1 week prior to the start of the intervention; (T3) Post-treatment: the week immediately following the intervention; (T4) Follow-up: 3 months after the conclusion of the intervention.
  Test of word retrieval and executive control abilities such as updating, shifting, and inhibiting. Participants are asked to name as many items as possible in 1 minute for a given category (e.g., clothes) and for a given letter (e.g., "s").
Change on the Philadelphia Naming Test (PNT) | (T1) Baseline: at the start of the study; (T2) Pre-treatment: 1 week prior to the start of the intervention; (T3) Post-treatment: the week immediately following the intervention; (T4) Follow-up: 3 months after the conclusion of the intervention.
  Aphasia naming test to assess word retrieval abilities. The score ranges from 0 to 100, with a higher score indicating greater naming ability.
Changes on the California Cognitive Assessment Battery (CCAB) | (T1) Baseline: at the start of the study; (T2) Pre-treatment: 1 week prior to the start of the intervention; (T3) Post-treatment: the week immediately following the intervention; (T4) Follow-up: 3 months after the conclusion of the intervention.
  This is a computerized assessment battery of cognitive tasks that provides a comprehensive assessment of different cognitive domains. These tasks include computerized version of standard cognitive tasks such as Trail making test, Stroop test, Digit and Spatial Span tasks, Verbal learning tasks. These tasks will require participants to memorize lists of words, digits, describe pictures, and draw on the tablet. Participant's verbal and pointing responses will be recorded. The following tasks will be used: BAVLT Encoding, Digit Span Forward, Digit Span Reverse, Picture Matching, Spatial Span, Finger Tapping, BAVLT Delayed Recall, Continuous Picture Naming, Picture Description, Simple Reaction Time, Trails A, Trails B, Stroop, Design Fluency, Picture Description Delayed Recall, Verbal Fluency.
Changes in Maximal Aerobic Capacity | (T1) Baseline: at the start of the study; (T2) Pre-treatment: 1 week prior to the start of the intervention; (T3) Post-treatment: the week immediately following the intervention.
  This is a measure of cardiorespiratory and metabolic fitness. Maximal Aerobic Capacity (VO2 Max) is the ability of the body to utilize oxygen to produce energy and is measured via a graded exercise test until volitional fatigue, while measuring consumption of oxygen with a computerized metabolic system. Typically measured on a treadmill, VO2 Max has also been found to be accurately and safely measured in stroke survivors on a recumbent stepper, which will be used in this study. A good VO2 Max varies greatly depending on age, and for older participants is typically between 30-40ml/kg/min (higher values indicate greater fitness).
Change on the 2-minute Step Test | (T1) Baseline: at the start of the study; (T2) Pre-treatment: 1 week prior to the start of the intervention; (T3) Post-treatment: the week immediately following the intervention; (T4) Follow-up: 3 months after the conclusion of the intervention.
  The number of knee raises completed in 2 minutes, raising each knee to a point midway between the patella (kneecap) and iliac crest (top hip bone)
Change on the 30-second chair stands | (T1) Baseline: at the start of the study; (T2) Pre-treatment: 1 week prior to the start of the intervention; (T3) Post-treatment: the week immediately following the intervention; (T4) Follow-up: 3 months after the conclusion of the intervention.
  The number of full stands from a seated position that can be completed in 30 seconds with arms folded across the chest.
Change on the Timed Up-and-Go Test | (T1) Baseline: at the start of the study; (T2) Pre-treatment: 1 week prior to the start of the intervention; (T3) Post-treatment: the week immediately following the intervention; (T4) Follow-up: 3 months after the conclusion of the intervention.
  The number of seconds it takes to get up from a seated position, walk 3 m, turn, and return to a seated position.
Change on the Functional Reach Test | (T1) Baseline: at the start of the study; (T2) Pre-treatment: 1 week prior to the start of the intervention; (T3) Post-treatment: the week immediately following the intervention; (T4) Follow-up: 3 months after the conclusion of the intervention.
  The number of inches reached forward with each arm with feet flat on the floor at hip width.
Change in Gait Speed | (T1) Baseline: at the start of the study; (T2) Pre-treatment: 1 week prior to the start of the intervention; (T3) Post-treatment: the week immediately following the intervention; (T4) Follow-up: 3 months after the conclusion of the intervention.
  The speed in meters per second for the middle 6 m of the 10 m walkway.

OTHER OUTCOMES:
Changes on the Narrative Discourse Sample | (T1) Baseline: at the start of the study; (T2) Pre-treatment: 1 week prior to the start of the intervention; (T3) Post-treatment: the week immediately following the intervention; (T4) Follow-up: 3 months after the conclusion of the intervention.
  Analysis of discourse samples elicited using the WAB-R picture description, the Cat rescue story and the Cinderella story retell, narrative tasks commonly used in aphasia research.
Changes on the Functional Gait Assessment (FGA) | (T1) Baseline: at the start of the study; (T2) Pre-treatment: 1 week prior to the start of the intervention; (T3) Post-treatment: the week immediately following the intervention; (T4) Follow-up: 3 months after the conclusion of the intervention.
  A multi-component assessment of postural stability during walking and ability to perform additional motor tasks while walking.
Change in Center for Epidemiological Studies Depression Scale (CES-D) | (T1) Baseline: at the start of the study; (T2) Pre-treatment: 1 week prior to the start of the intervention; (T3) Post-treatment: the week immediately following the intervention; (T4) Follow-up: 3 months after the conclusion of the intervention.
  The 20-item self-rating questionnaire evaluates perceived mood and level of functioning within the past seven days. The scores range from 0-60. A score equal to or above 16 indicates a person at risk for clinical depression.
Changes on the General Anxiety Disorder scale (GAD-7) | (T1) Baseline: at the start of the study; (T2) Pre-treatment: 1 week prior to the start of the intervention; (T3) Post-treatment: the week immediately following the intervention; (T4) Follow-up: 3 months after the conclusion of the intervention.
  The 7-item self-report scale is used to identify anxiety based on problems experienced in the last two weeks. The scores range from 0-21, with higher scores indicative of more pronounced anxiety symptoms.
Changes on the Pittsburgh Sleep Quality Index (PSQI) | (T1) Baseline: at the start of the study; (T2) Pre-treatment: 1 week prior to the start of the intervention; (T3) Post-treatment: the week immediately following the intervention; (T4) Follow-up: 3 months after the conclusion of the intervention.
  The self-rating scale used to measure the quality and patterns of sleep. It differentiates "poor" from "good" sleep by measuring seven areas: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction over the last month. The overall score ranges from 0-21, with higher scores indicative of more acute sleep disturbances.
Changes on the Stroke and Aphasia Quality of Life Scale - 39 (SAQOL-39) | (T1) Baseline: at the start of the study; (T2) Pre-treatment: 1 week prior to the start of the intervention; (T3) Post-treatment: the week immediately following the intervention; (T4) Follow-up: 3 months after the conclusion of the intervention.
  This questionnaire is specifically designed to assess quality of life in individuals with stroke and aphasia. The overall quality of life score can range from 1 to 5, with higher values indicating better quality of life and overall well-being.
Changes on the Fugl-Meyer Assessment, Upper Extremity portion (FMA-UE) | (T1) Baseline: at the start of the study or (T2) Pre-treatment: 1 week prior to the start of the intervention; (T3) Post-treatment: the week immediately following the intervention.
  This is a commonly used outcome measure for assessment of sensorimotor recovery after stroke. We will only use the upper extremity portion of the assessment to supplement other study measures focusing on gait and balance. The FMA-UE assesses movement, coordination, and reflexes associated with the shoulder, elbow, forearm, wrist, and hand and is meant to capture stages of motor recovery after stroke. The FMA-UE consists of 33 items with each item scored on a 3-point ordinal scale (0, 1, or 2), with 0 generally corresponding to no function, 1 to partial function, and 2 to perfect function. The items are summed to provide a final score, ranging from 0-66 points, with lower scores indicative of more pronounced motor impairments of the upper extremity.
Change on the Modified Rankin Scale (MRS) | (T1) Baseline: at the start of the study or (T2) Pre-treatment: 1 week prior to the start of the intervention; (T3) Post-treatment: the week immediately following the intervention.
  This is a commonly used 7-point rating scale for measuring the degree of overall disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. MRS is a single item, global outcomes rating scale for patients post-stroke. The measure is scored based on a structured interview. It is used to categorize level of functional independence with reference to pre-stroke activities rather than on observed performance of a specific task. The scale ranges from 0 to 6, with higher scores indicative of more severe disability, with 6 indicating that the patient is dead.
Changes on the National Institute of Health Stroke Scale (NIHSS) | (T1) Baseline: at the start of the study or (T2) Pre-treatment: 1 week prior to the start of the intervention; (T3) Post-treatment: the week immediately following the intervention.
  This is a widely used clinical scale for measuring impairment in various domains (consciousness, motor, sensory, attention, language) after stroke. It uses a numerical scale to determine stroke severity, health care providers record the person's performance in 11 categories, such as sensory and motor ability. Each domain is rated on a scale from 0 to 2 or3/4 for certain domains), with 0 indicating no impairment. The total score can range from 0 to 42 points, with higher scores indicating greater severity.
Change in blood pressure at rest | (T1) Baseline: at the start of the study; (T2) Pre-treatment: 1 week prior to the start of the intervention; (T3) Post-treatment: the week immediately following the intervention.
  Both systolic and diastolic blood pressure will be measured at rest with a manual blood pressure monitor.
Change in Stepping Cadence | Two one-week periods: one week prior to and one week following the intervention.
  To evaluate overall daily activity levels in the real world, physical activity and sedentary behavior will be recorded using the activPAL4+ activity monitor (PAL Technologies Ltd., Glasgow, UK). The activPAL is a research-grade device that uses a combination of an accelerometer, inclinometer, and gyroscope to objectively measure time spent in different postures, including lying, sitting, standing, and stepping, as well as the intensity and duration of physical activity. We will track the following outcomes to evaluate changes in stepping cadence: steps per day, steps per minute (cadence), and peak 30-minute cadence.
Change in Activity Levels | Two one-week periods: one week prior to and one week following the intervention.
  To evaluate overall daily activity levels in the real world, physical activity and sedentary behavior will be recorded using the activPAL4+ activity monitor (PAL Technologies Ltd., Glasgow, UK). The activPAL is a research-grade device that uses a combination of an accelerometer, inclinometer, and gyroscope to objectively measure time spent in different postures, including lying, sitting, standing, and stepping, as well as the intensity and duration of physical activity. We will track the following outcomes to evaluate changes in activity levels: standing time (in minutes), sitting time (in minutes), lying time (in minutes), number of sit-to-stand transitions, lying bouts greater than 30 minutes, and stepping bouts greater than 5 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Maria Ivanova, PhD, Principal Investigator — University of California, Berkeley
Locations (4):
- United States (4):
  - University of California, Berkeley, Berkeley, California
  - California State University, East Bay, Hayward, California
  - University of San Francisco, San Francisco, California
  - University of California, San Francisco, San Francisco, California

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication

REFERENCES:
- See also: Related Info — https://apex.berkeley.edu/